CLINICAL TRIAL: NCT03272230
Title: Assessment of Apathy in a Real-life Situation, With a Video and Sensors-based System in Healthy Subject and Patient With Cerebral Disease
Brief Title: Assessment of Apathy in a Real-life Situation, With a Video and Sensors-based System
Acronym: ECOCAPTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Brain Institute Paris (ICM) (Unknown); Pitié-Salpêtrière Hospital (AP-HP) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C16-87; 2017-A00416-47 (Registry Identifier: RCB)
Record Dates: First submitted 2017-08-03; First posted 2017-09-05 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Apathy; Behavioral Variant Frontotemporal Dementia (bvFTD); Disinhibition; Depression - Major Depressive Disorder
Keywords: Apathy; Goal-directed behavior; Assessment; Diagnosis; Sensor; Ecological condition; Neurological disease; Dementia; Human ethology; Behavioral sensing; Accelerometer; Disinhibition; ECOCAPTURE
MeSH Terms: conditions — Lethargy; Disease; Nervous System Diseases; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): The Arm consists of two separate visits, each occurring on a different day, and includes the following components: the ECOCAPTURE observation phase in ecological conditions, a comprehensive neuropsychological assessment, a series of experimental tasks (some of which are computer-based), an MRI scan (including T1, T2, rs-fMRI, and MS-DWI), and a blood sample collection.
  Interventions: Behavioral: ECOCAPTURE; Behavioral: Cognitive and Behavioral experimental tasks; Diagnostic Test: Neuropsychological assessment; Behavioral: ICM_APATHY_TASKS; Other: MRI; Biological: Neurohormonal mechanisms

INTERVENTIONS:
Behavioral: ECOCAPTURE — 45 minutes observational session for tracking goal directed behavior into a waiting room equipped with video and sensor-based data acquisition system
Behavioral: Cognitive and Behavioral experimental tasks — Cognitive and Behavioral experimental tasks to explore additional frontal cognitive and behavioral dimensions and functions
Diagnostic Test: Neuropsychological assessment — STARKSTEIN APATHY SCALE (SAS) / DAS / MMSE / MADRS / EBI / MINI-SEA / FAB / HAD / MATTIS / HAYLING / STROOP / Verbal Span / Lexical verbal fluency / TMT / CDRS
Behavioral: ICM_APATHY_TASKS — Apathy experimental task
Other: MRI — T1 / T2 / rs-fMRI / MS-DWI
Biological: Neurohormonal mechanisms — Hormonal dosage / Diabetic dosage / Ionogramme dosage / Inflammatory dosage / Hepatic dosage / Lipidic dosage / Thyroid dosage

SUMMARY:
Apathy is defined as a quantitative reduction in voluntary and goal-directed behavior. To address this, the investigators propose an ethological approach to assess apathy objectively and quantitatively by observing patients in real-life situations.

The ECOCAPTURE paradigm involves a structured, multi-step scenario conducted in a functional exploration platform. This platform is equipped with an advanced data acquisition system integrating video recordings and sensors to precisely monitor and analyze participants' behavior.

Primary objective:

Develop a diagnostic tool for apathy using metrics derived from video recordings and sensor data. This tool aims to provide objective measures to identify and quantify apathy.

Secondary Objectives:

* Validation of ICM_APATHY_TASKS: This novel experimental task is designed to evaluate three primary mechanisms thought to underlie apathy: Motivation, Cognitive inertia (difficulty initiating tasks), The interaction between motivation and action execution.
* Identification of the pathophysiological mechanisms of apathy by investigate the cognitive, behavioral, neural, and neurohormonal underpinnings of apathy.

This will enable the classification of apathetic patients into subtypes (or several forms of apathy) based on the dominant mechanisms and provide insights into which processes best explain apathy in individual cases.

This innovative framework aims to deepen the understanding of apathy, improve diagnostic precision, and pave the way for tailored interventions.

DETAILED DESCRIPTION:
A pilot study, ECOCAPTURE (ClinicalTrials.gov/NCT02496312, 2015), was conducted with participants diagnosed with the behavioral variant of frontotemporal dementia (bvFTD) matched for age, gender, and education level with healthy controls (n=7 per group). This study successfully validated the feasibility and conceptual framework of the ECOCAPTURE approach.

The aim of this trial is to further develop and expand the ECOCAPTURE tool by applying it to a larger population, including individuals with the behavioral variant of frontotemporal dementia (bvFTD) and healthy control participants.

The objectives of this study are to evaluate goal-directed behavior and identify apathy by analyzing data to establish a behavioral signature of apathy. Additionally, the study seeks to refine patient profiles by delineating the pathophysiological mechanisms underlying apathy, including cognitive processes, neural substrates, and neurohormonal pathways.

The experiments take place on an experimental platform dedicated to the functional exploration of human behavior (PRISME, ICM core facility, Salpêtrière Hospital, Paris, France), to assess behavior under ecological conditions. The ECOCAPTURE paradigm mimics a naturalistic situation (i.e., waiting comfortably in a waiting room). Participants undergo a structured 45-minute controlled scenario, during which their behavior is systematically monitored to evaluate apathy and disinhibition.

The PRISME platform is transformed into a furnished waiting room containing specific objects that provides opportunities to interact with the environment. The platform is equipped with a six-ceiling camera system (not hidden) covering the entire waiting room. The Media Recorder® software (NOLDUS Information Technology, Wageningen, the Netherlands) facilitates simultaneous video recordings from multiple cameras, ensuring synchronized capture across different viewpoints for comprehensive behavioral analysis. During the experiment, individuals' behavior is video-recorded, and their movement acceleration is measured using a wireless body sensor (Move II® triaxial accelerometer, Movisens GmbH, Karlsruhe, Germany) worn on the right hip. An eye-tracking system (SMI Eye Tracking Glasses 2 Wireless, ®SensoMotoric Instruments, Teltow, Germany / Tobii Pro Glasses 3, ®Tobii AB, Danderyd, Sweden) is added to the multimodal recording system, and the subjects wear eye-tracking glasses for a 7-minute period during the 45-minute experimental session. The subjects are informed at the time of initial consent that their behavior would be tracked and recorded by video cameras located in the room.

Video data analysis is performed with The Observer XT software (Version 14.0, NOLDUS, Wageningen, The Netherlands) to identify the frequency and duration of behaviors. Behavioral metrics are obtained by behavioral coding from 45-minute video footage for each individual. Behavioral coding data is collected through the continuous sampling method, to identify all occurrences of behaviors and their duration. Behavioral coding is conducted based on two ethograms - the ECOCAPTURE apathy ethogram, the ECOCAPTURE disinhibition ethogram - (Batrancourt et al. 2022, "The ECOCAPTURE ethograms: apathy ethogram and disinhibition ethogram", Mendeley Data, V2, doi: 10.17632/mv8hndcd95.2) The ECOCAPTURE apathy ethogram includes behaviors divided in two behavioral categories: Motor patterns, Activity states. The ECOCAPTURE disinhibition ethogram includes behaviors divided in three disinhibition categories: Compulsivity, Impulsivity, Social disinhibition.

Metrics built from collected data (video, sensors) are analyzed to reveal a behavioral signature of apathy.

The study consists of two separate visits, each occurring on a different day, and includes the following components: the ECOCAPTURE observation phase in ecological conditions, a comprehensive neuropsychological assessment, a series of experimental tasks (some of which are computer-based), an MRI scan (including T1, T2, rs-fMRI, and MS-DWI), and a blood sample collection.

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria for All Groups:

* Demonstrates the ability to provide informed consent for participation in the study.
* Capable of understanding study instructions and performing cognitive tasks as required.
* Enrolled in a valid health insurance plan.

Eligibility Criteria for Patients:

* Mini-Mental State Examination (MMSE): Score ≥ 17.
* Medical History: Absence of any other neurological or psychiatric conditions.
* Caregiver Requirement: Must have a caregiver present.

Patient Groups:

* Diagnosed with behavioral variant frontotemporal dementia (bvFTD) based on the Rascovsky criteria (Rascovsky et al., 2011).
* Diagnosed with Major Depressive Disorder (MDD) according to DSM-IV criteria.

Eligibility Criteria for Healthy Age-, Sex-, and Education-Matched Controls:

* Mini-Mental State Examination (MMSE): Score > 27.
* Medical History: No history of neurological or psychiatric disorders.

Exclusion Criteria:

* MRI Contraindications: Standard contraindications to magnetic resonance imaging (e.g., pacemaker, metallic implants, claustrophobia).
* Cognitive Barriers: Inability to comprehend study instructions.
* Legal Restrictions: Individuals referenced in Articles L.1121-5 to L.1121-8 and L.1122-12 of the French Public Health Code.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Frequency of each behavior in the ECOCAPTURE ethogram | 45 min
  [Tracking specific behaviors as outlined in the ECOCAPTURE ethogram. Behavioral metrics are derived from coding the behaviors observed in 45-minute video footage, based on the structured ethogram] integer.
  .
Occurrence of each behavior in the ECOCAPTURE ethogram | 45 min
  [Tracking specific behaviors as outlined in the ECOCAPTURE ethogram. Behavioral metrics are derived from coding the behaviors observed in 45-minute video footage, based on the structured ethogram] integer.
  .
Duration of each behavior in the ECOCAPTURE ethogram | 45 min
  [Tracking specific behaviors as outlined in the ECOCAPTURE ethogram. Behavioral metrics are derived from coding the behaviors observed in 45-minute video footage, based on the structured ethogram] integer.
  .
Activity classes | 45 min
  [Provided by the accelerometer sensor] Activity class: Indicates the physical position of the subject (unknown position = 0, lying down = 1, sitting/standing = 2, vertical movement upwards = 4, fast movement = 5, vertical movement downwards = 6, walking = 7)
Body positions | 45 min
  [Provided by the accelerometer sensor] Body position: Specifies the characteristics of the lying position (unknown position = 0, lying on the back = 1, lying on the left side = 2, lying on the stomach = 3, lying on the right side = 4, getting up = 5).
Steps | 45 min
  [Provided by the accelerometer sensor] Counting steps.
Energy expenditure | 45 min
  [Provided by the accelerometer sensor] Energy expenditure during activity phases. kcal.
MET | 45 min
  [Provided by the accelerometer sensor] The Metabolic Equivalent of Task: MET level.
Acceleration intensity | 45 min
  [Provided by the accelerometer sensor] g.
Pupil Diameter x,y | 7 min
  [Provided by the eye-tracking glasses] mm, mm.
Ocular events | 7 mn
  [Provided by the eye-tracking glasses] Saccades, Fixations and Blink frequency.
Gaze points | 7 mn
  [Provided by the eye-tracking glasses] Individual records of the participant's gaze at any given moment

SECONDARY OUTCOMES:
STARKSTEIN (SAS) | 10 mn
  [Part of the neuropsychological assessment - Starkstein Apathy Scale] SAS global score
DAS | 10 mn
  [Part of the neuropsychological assessment] - Dimensional Apathy Scale - DAS global score - DAS initiation score - DAS executive score - DAS emotional score.
ICM_APATHY_TASKS | 1 hour
  ICM_APATHY_TASKS global score. [The ICM_APATHY_TASKS test three main presumed mechanisms of apathy: lack of motivation, cognitive inertia, and the decoupling between motivation and action. These tasks integrate two orthogonal dimensions: 1/ The cognitive dimension: modulation of the level of cognitive strategy (to study cognitive inertia); 2/ The motivational dimension: modulation of the reward at stake (to study lack of motivation)].
MMSE | 5 mn
  [Part of the neuropsychological assessment] - Mini Mental State Exam - MMSE global score
MADRS | 10 mn
  [Part of the neuropsychological assessment] - Montgomery-Åsberg Depression Rating Scale - MADRS global score
EBI | 15 mn
  [Part of the neuropsychological assessment] - Eating Behavior Inventory - EBI scores. [Food behavior questionnaire. This refers to an assessment tool designed to evaluate a person's eating behaviors and identify potential risks, such as choking or aspiration, during eating].
MATTIS | 20 mn
  [Part of the neuropsychological assessment] - Mattis Dementia Rating Scale - MATTIS global score
FAB | 10 mn
  [Part of the neuropsychological assessment] - Frontal Assessment Battery - FAB global score [French version: BREF].
HAYLING | 15 mn
  [Part of the neuropsychological assessment] - Hayling Sentence Completion test - HAYLING B-A score
HAD | 10 mn
  [Part of the neuropsychological assessment] Hospital Anxiety and Depression Scale - HAD global score
STROOP | 3 mn
  [Part of the neuropsychological assessment] - STROOP - STROOP global score
Mini-SEA | 20 mn
  [Part of the neuropsychological assessment] - Mini Social cognition and Emotional Assesment - Mini-SEA global score
Verbal Span / Lexical verbal fluency | 7 mn
  [Part of the neuropsychological assessment] - Verbal Span / Lexical verbal fluency - Verbal scores
CDRS | 5 mn
  [Part of the neuropsychological assessment] - Clinical Dementia Rating (CDR) Scale - CDRS global score
Gray matter volume | MRI exam: 48 mn
  [MRI analysis- Brain segmentation] mm3
White matter volume | MRI exam: 48 mn
  [MRI analysis- Brain segmentation] mm3
Cortical Thickness | MRI exam: 48 mn
  [MRI analysis- Brain segmentation] mm
Resting-State Connectivity | MRI exam: 48 mn
  [fMRI analysis] - strength and significance of the connection between different regions.
IL-6 | Blood sample collection - 30 mn
  Hormonal result [Interleukin-6] pg/mL
Leptin | Blood sample collection - 30 mn
  Hormonal result [Leptin] ng/mL
Adiponectin | Blood sample collection - 30 mn
  Hormonal result [Blood adiponectin level)] mg/L
Insulin | Blood sample collection - 30 mn
  Hormonal result [Fasting Insulin] mUI/L
C-Peptide | Blood sample collection - 30 mn
  Diabetic result [Fasting C-Peptide level] µg/L
FPG | Blood sample collection - 30 mn
  Diabetic result [Fasting Plasma Glucose] mmol/L
HbA1C | Blood sample collection - 30 mn
  Diabetic result [Glycated Hemoglobin] %
Sodium | Blood sample collection - 30 mn
  Ionogram result [Sodium] mmol/L
K+ | Blood sample collection - 30 mn
  Ionogram result [Potassium] mmol/L
Uric acid | Blood sample collection - 30 mn
  Ionogram result [Uric acid] µmol/L
Creatinine | Blood sample collection - 30 mn
  Ionogram result [Creatinine] µmol/L
Total Protein | Blood sample collection - 30 mn
  Ionogram result [Total protein] g/L
CRP | Blood sample collection - 30 mn
  Inflammatory result [C-reactive protein] mG/L
AST | Blood sample collection - 30 mn
  Hepatic result [Aspartate aminotransferase] U/L
ALT | Blood sample collection - 30 mn
  Hepatic result [Alanine aminotransferase] U/L
GGT | Blood sample collection - 30 mn
  Hepatic result [Gamma-glutamyltransferase] U/L
Cholesterol | Blood sample collection - 30 mn
  Lipidic result [Total cholesterol] mmol/L
Triglycerides | Blood sample collection - 30 mn
  Lipidic result [Triglycerides] mmol/L
HDL cholesterol | Blood sample collection - 30 mn
  Lipidic result [High-density lipoprotein cholesterol] mmol/L
LDL cholesterol | Blood sample collection - 30 mn
  Lipidic result [Low-density lipoprotein cholesterol] mmol/L
Glycerol | Blood sample collection - 30 mn
  Lipidic result [Plasma glycerol concentration] mmol/L
FFAs | Blood sample collection - 30 mn
  Lipidic result [Plasma free fatty acids] mmol/L
TSH | Blood sample collection - 30 mn
  Thyroid result [Thyroid-stimulating hormone blood test] mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Richard LEVY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Bénédicte BATRANCOURT, PhD, Study Chair — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Paris Brain Institute / ICM / Pitié-Salpêtrière Hospital AP-HP / CIC, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The scientific leaders of the ECOCAPTURE research project aim to participate in international OPEN DATA initiatives. In this context, the following fully anonymized data will be made available to the scientific community:
  * Data collected from the accelerometer-type sensor.
  * Data on the subject's ocular behavior (events such as saccades or fixations) from the eye-tracking sensor. The videos from the glasses will not be shared.
  * Behavioral data from video coding based on the ECOCAPTURE ethogram. The videos will not be shared.
  * Scores from the neuropsychological assessment
  * MRI data
  * Blood test data.
Supporting Information: Study Protocol
Time Frame: 2026-2030
Access Criteria: Researchers must contact the scientific leaders of the study, and an agreement must be established with the sponsor (INSERM).

REFERENCES:
- [Result] Godefroy V, Tanguy D, Bouzigues A, Sezer I, Ferrand-Verdejo J, Azuar C, Bendetowicz D, Carle G, Rametti-Lacroux A, Bombois S, Cognat E, Jannin P, Morandi X, Ber IL, Levy R, Batrancourt B, Migliaccio R. Frontotemporal dementia subtypes based on behavioral inhibition deficits. Alzheimers Dement (Amst). 2021 Apr 6;13(1):e12178. doi: 10.1002/dad2.12178. eCollection 2021. PMID 33851004
- [Result] Godefroy V, Batrancourt B, Charron S, Bouzigues A, Bendetowicz D, Carle G, Rametti-Lacroux A, Bombois S, Cognat E, Migliaccio R, Levy R. Functional connectivity correlates of reduced goal-directed behaviors in behavioural variant frontotemporal dementia. Brain Struct Funct. 2022 Dec;227(9):2971-2989. doi: 10.1007/s00429-022-02519-5. Epub 2022 Jun 25. PMID 35751676
- [Result] Godefroy V, Batrancourt B, Charron S, Bouzigues A, Sezer I, Bendetowicz D, Carle G, Rametti-Lacroux A, Bombois S, Cognat E, Migliaccio R, Levy R. Disentangling Clinical Profiles of Apathy in Behavioral Variant Frontotemporal Dementia. J Alzheimers Dis. 2022;90(2):639-654. doi: 10.3233/JAD-220370. PMID 36155506
- [Result] Godefroy V, Durand A, Simon MC, Weber B, Kable J, Lerman C, Bergstrom F, Levy R, Batrancourt B, Schmidt L, Plassmann H, Koban L. A structural MRI marker predicts individual differences in impulsivity and classifies patients with behavioral-variant frontotemporal dementia from matched controls. bioRxiv [Preprint]. 2024 Sep 16:2024.09.12.612706. doi: 10.1101/2024.09.12.612706. PMID 39345385
- [Result] Batrancourt B, Lecouturier K, Ferrand-Verdejo J, Guillemot V, Azuar C, Bendetowicz D, Migliaccio R, Rametti-Lacroux A, Dubois B, Levy R. Exploration Deficits Under Ecological Conditions as a Marker of Apathy in Frontotemporal Dementia. Front Neurol. 2019 Aug 28;10:941. doi: 10.3389/fneur.2019.00941. eCollection 2019. PMID 31551908
- [Result] Peltier C, Lejeune FX, Jorgensen LGT, Rametti-Lacroux A, Tanguy D, Godefroy V, Bendetowicz D, Carle G, Cognat E, Bombois S, Migliaccio R, Levy R, Marin F, Batrancourt B; ECOCAPTURE study group. A temporal classification method based on behavior time series data in patients with behavioral variant of frontotemporal dementia and apathy. J Neurosci Methods. 2022 Jul 1;376:109625. doi: 10.1016/j.jneumeth.2022.109625. Epub 2022 May 30. PMID 35653896
- [Result] Tanguy D, Batrancourt B, Estudillo-Romero A, Baxter JSH, Le Ber I, Bouzigues A, Godefroy V, Funkiewiez A, Chamayou C, Volle E, Saracino D, Rametti-Lacroux A, Morandi X, Jannin P, Levy R, Migliaccio R; ECOCAPTURE study group. An ecological approach to identify distinct neural correlates of disinhibition in frontotemporal dementia. Neuroimage Clin. 2022;35:103079. doi: 10.1016/j.nicl.2022.103079. Epub 2022 Jun 7. PMID 35700600
- [Result] Tanguy D, Rametti-Lacroux A, Bouzigues A, Saracino D, Le Ber I, Godefroy V, Morandi X, Jannin P, Levy R, Batrancourt B, Migliaccio R; ECOCAPTURE Study Group. Behavioural disinhibition in frontotemporal dementia investigated within an ecological framework. Cortex. 2023 Mar;160:152-166. doi: 10.1016/j.cortex.2022.11.013. Epub 2022 Dec 28. PMID 36658040
- Available data/document: Study Protocol — https://data.mendeley.com/datasets/mv8hndcd95/2 — The ECOCAPTURE ethograms: apathy ethogram and disinhibition ethogram
- Available data/document: Individual Participant Data Set — https://data.mendeley.com/datasets/vdrstwp5xx/1 — ECOCAPTURE Dataset - Behavioral coding from video - 17 bvFTD and 18 HC - 28.04.2022
- Available data/document: Individual Participant Data Set — https://data.mendeley.com/datasets/p88gtz8wdz/4 — ECOCAPTURE Dataset - Behavioral coding from video - 20 bvFTD and 18 HC - 21.03.2022
- Available data/document: Individual Participant Data Set — https://data.mendeley.com/datasets/6n7p3y3j58/2 — ECOCAPTURE Dataset - Behavioral coding from video - 23 bvFTD and 24 HC - 28.11.2022